CLINICAL TRIAL: NCT00945789
Title: Human Recombinant Erythropoietin (HrEPO) in Asphyxia Neonatorum: A Pilot Trial
Brief Title: Erythropoietin in Infants With Hypoxic Ischemic Encephalopathy (HIE)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Abdul rahman Al Mashad, MD Associate Professor of Pediatrics, Tanta University Faculty of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1102007
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Last update posted 2009-09-28 (Estimated); Status verified 2009-09

CONDITIONS: Hypoxic Ischemic Encephalopathy
Keywords: Asphyxia neonatorum; Infants; EEG; Brain MRI; Nitric oxide
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Asphyxia Neonatorum | interventions — Endothelium-Dependent Relaxing Factors

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- EPO HIE Group (Experimental): Infants with hypoxic ischemic encephalopathy receive human recombinant erythropoietin
  Interventions: Drug: Human recombinant erythropoietin; Procedure: EEG and Brain MRI; Biological: Nitric oxide measurement in the blood
- Control HIE (No Intervention): Infants with hypoxic ischemic encephalopathy who do not receive treatment drug (EPO)
  Interventions: Procedure: EEG and Brain MRI; Biological: Nitric oxide measurement in the blood
- Healthy Controls (Other): Healthy newborn without hypoxic ischemic encephalopathy
  Interventions: Biological: Nitric oxide measurement in the blood

INTERVENTIONS:
Drug: Human recombinant erythropoietin — Epo dse is 2500 IU/kg subcutaneous daily for 5 days.
  Arms: EPO HIE Group
Procedure: EEG and Brain MRI — EEG to be done twice in hte first 48 hours and at 2-3 weeks. MRI to be done at 3 weeks of age.
  Arms: Control HIE; EPO HIE Group
Biological: Nitric oxide measurement in the blood — Concentration of nitric oxide is measured in the blood at enrollment. For the 2 groups with asphyxia, measurement to be repeated in 2 weeks.

SUMMARY:
In this prospective trial the investigators plan to study the efficacy of erythropoietin as a therapeutic agent in neonates who suffer from brain injury following perinatal asphyxia.

DETAILED DESCRIPTION:
During HIE free radicals are generated within mitochondria and also as byproducts in the synthesis of prostaglandins.These free radicals ignite a secondary phase of subsequent damage to the brain by attacking membranal fatty acids. Nitric oxide (NO) is involved in the cascade of metabolic events that contributes to HIE. It mediates, in part, the cytotoxic activity of macrophages, induces relaxation of blood vessels, and also acts as a neurotransmitter in the central and peripheral nervous system. Therefore, the therapeutic value of NO synthase inhibitors, among many other agents used to ameliorate the course of HIE, is currently under investigation in experimental animals.

Erythropoietin (EPO) is a cytokine originally identified for its role in erythropoiesis and more recently shown to be produced in the central nervous system.Relative insufficiency of endogenous EPO during periods of ischemic stress may trigger neuronal apoptosis, whereas the provision of exogenous EPO has been shown to inhibit this process. The potential immediate protective effects of EPO include decreased NO production, activation of antioxidant enzymes, reduction of glutamate toxicity, inhibition of lipid peroxidation, and reduction of inflammation. Long-term protective effects of EPO include the generation of neuronal anti-apoptotic mechanisms, stimulation of angiogenesis, and modulation of neurogenesis.

Preliminary data supports a protective role of exogenous EPO to neuronal cells. The presence of EPO rescues in vitro cultured neurons from NO-induced death. It specifically protects cultured neurons from N-methyl-D-aspartate (NMDA) receptor-mediated glutamate toxicity. Intercerebroventricular injection of EPO offered significant protection of neuronal tissue in animals with focal cerebral ischemia. EPO is able to cross the blood brain barrier, and its concentration in the cerebrospinal fluid in normal rats significantly increases within 30 minutes following intravenous administration. EPO also offered neuronal protection when it was administered systemically to animals suffering from global and focal cerebral ischemia. In adult patients with stroke, the administration of EPO ameliorates the course of the disease. Therefore, EPO has recently received much attention and is speculated to have a role in the protection of HIE infants. However, despite the biological plausibility and the encouraging preliminary data from animals and adult humans, surprisingly EPO has never been tried in newborns with HIE even though it has already been used in neonates for other indications and is known to be safe.

ELIGIBILITY:
Inclusion Criteria:

* Inborn infants at term gestation (38-42 weeks)
* Apgar score ≤ 3 at 5 minutes and/or delayed first breath beyond five minutes after birth
* Profound metabolic or mixed acidosis with serum bicarbonate <12 mMol/L in initial arterial blood gas
* Evidence of encephalopathy such as stupor, coma, seizures, or hypotonia in the immediate neonatal period

Exclusion Criteria:

* Twin gestation
* Maternal diabetes
* Congenital malformations of the central nervous system
* Chromosomal abnormalities
* Chorioamnionitis and congenital infections
* Intrauterine growth restriction

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2007-10; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Neurodevelopmental outcomes | 6 months
EEG changes | 2-3 weeks
MRI of the brain | 3 weeks

SECONDARY OUTCOMES:
Nitric oxide concentrations in the plasma | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Faculty of Medicine, Tanta, Egypt

REFERENCES:
- [Derived] Elmahdy H, El-Mashad AR, El-Bahrawy H, El-Gohary T, El-Barbary A, Aly H. Human recombinant erythropoietin in asphyxia neonatorum: pilot trial. Pediatrics. 2010 May;125(5):e1135-42. doi: 10.1542/peds.2009-2268. Epub 2010 Apr 12. PMID 20385632